CLINICAL TRIAL: NCT04294771
Title: JOint Use of Database to Identify Risk Factors of CARDio-vascular Adverse Reactions Induced by Immune Checkpoint InhibiTors: VigiBase, Entrepot de Données de Santé (EDS), Système National Des Données de Santé (SNDS) Databases and a Retrospective International Multicenter Registry of ICI-associated Myocarditis
Brief Title: JOint Use of Database to Identify Risk Factors of CARDio-vascular Toxicity Induced by Immune Checkpoint Inhibitors
Acronym: JOCARDITE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, Principal Investigator, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-20-03
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Myocarditis; Cardiomyopathies; Heart Diseases; Cardiovascular Diseases; Pericarditis; Vasculitis
Keywords: Drug-induced cardiotoxicity; Immune Checkpoint Inhibitors; Anti-PD-1; Anti-PD-L1; Anti CTLA-4
MeSH Terms: conditions — Myocarditis; Cardiomyopathies; Heart Diseases; Cardiovascular Diseases; Pericarditis; Vasculitis | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Myocarditis and other cardiovascular toxicities ICI-related: Case reported in the World Health Organization (WHO)international pharmacovigilance database, or APHP Entrepot de Données de Santé (EDS) and French Système National Des Données de Santé (SNDS) Databases, with a chronology compatible with the drug toxicity
  Interventions: Drug: ICI
- Non case: Non-case will be patients exposed to ICI without cardiovascular toxicities
  Interventions: Drug: ICI

INTERVENTIONS:
Drug: ICI — Immune checkpoint inhibitor targeting either PD-1, PD-L1 or CTLA-4, and included in the ATC following list (ATC classification): Ipilimumab (L01XC11), Nivolumab (L01XC17), Pembrolizumab (L01XC18), Durvalumab (L01XC28), Avelumab (L01XC31), Atezolizumab (L01XC3)
  Other Names: Immune checkpoint inhibitors

SUMMARY:
Immune checkpoint inhibitors (ICIs) might induce high grade immune-related adverse events (irAEs) involving the cardio-vascular system. This study investigates reports of cardio-vascular toxicity associated with treatment including anti-PD1, Anti-PDL-1, and Anti CTLA4 classes using the World Health Organization (WHO) database VigiBase, Assistance Publique Hopitaux de Paris Entrepot de Données de Santé (APHP.EDS), French Système National Des Données de Santé (SNDS) Databases and a retrospective international multicenter registry of ICI-associated myocarditis

DETAILED DESCRIPTION:
ICIs have dramatically improved clinical outcomes in multiple cancer types and are increasingly being tested in earlier disease settings and in combination. Thus, irAEs can occur and risk factors for such events have been scarcely described. Here, the investigators will use VigiBase (http://www.vigiaccess.org/), the World Health Organization (WHO) database of individual safety case reports, to identify risk factors for cases of cardiovascular adverse drug reaction following treatment with ICIs, the investigators will also use two french databases : APHP Entrepot de Données de Santé (EDS), French Système National Des Données de Santé (SNDS) Databases and a retrospective international multicenter registry of ICI-associated myocarditis

ELIGIBILITY:
Inclusion Criteria:

* Case reported in the World Health Organization (WHO) database of individual safety case reports to 01/01/2025
* Case reported in the APHP Entrepot de Données de Santé (EDS) database of individual safety case reports to 01/01/2025
* Case reported in the Système National Des Données de Santé (SNDS) Database of individual safety case reports to 01/01/2025
* Case reported in a retrospective international multicenter registry of ICI-associated myocarditis to 01/01/2025
* Adverse event reported were including the MedDRA terms: Cardiac and vascular investigations (excl enzyme tests) (HLGT), Vascular disorders (SOC), Skeletal and cardiac muscle analyses (HLT), Sudden death (PT), Sudden cardiac death (PT), Cardiac disorders (SOC), Cardiac arrhythmias (HLGT), Cardiac disorder signs and symptoms (HLGT), Cardiac neoplasms (HLGT), Cardiac valve disorders (HLGT), Congenital cardiac disorders (HLGT), Coronary artery disorders (HLGT), Endocardial disorders (HLGT), Heart failures (HLGT), Myocardial disorders (HLGT), Pericardial disorders (HLGT)
* Patients treated with ICIs included in the ATC: Ipilimumab (L01XC11), Nivolumab (L01XC17), Pembrolizumab (L01XC18), Durvalumab (L01XC28), Avelumab (L01XC31), Atezolizumab (L01XC32), Cemiplimab (L01XC33)

Exclusion Criteria:

* Chronology not compatible between the drug and the toxicity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with an ICI for a cancer
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Identifying risk factors of cardio-vascular toxicity of ICIs. | Case reported in VigiBase, APHP Entrepot de Données de Santé (EDS), Système National Des Données de Santé (SNDS) Databases and a retrospective international multicenter registry of ICI-associated myocarditis from inception to January 2025
  Identifying risk factors of overreporting of cardiovascular adverse events in ICI treated patients

SECONDARY OUTCOMES:
Causality assessment of reported cardiovascular events | Case reported in VigiBase, APHP Entrepot de Données de Santé (EDS), Système National Des Données de Santé (SNDS) Databases and a retrospective international multicenter registry of ICI-associated myocarditis from inception to January 2025
Description of the type of cardiotoxicity depending on the category of ICIs | Case reported in VigiBase, APHP Entrepot de Données de Santé (EDS), Système National Des Données de Santé (SNDS) Databases and a retrospective international multicenter registry of ICI-associated myocarditis from inception to January 2025
Description of the duration of treatment when the toxicity happens (role of cumulative dose) | Case reported in VigiBase, APHP Entrepot de Données de Santé (EDS), Système National Des Données de Santé (SNDS) Databases and a retrospective international multicenter registry of ICI-associated myocarditis from inception to January 2025
Description of the drug-drug interactions associated with adverse events | Case reported in VigiBase, APHP Entrepot de Données de Santé (EDS), Système National Des Données de Santé (SNDS) Databases and a retrospective international multicenter registry of ICI-associated myocarditis from inception to January 2025
Description of the pathologies (cancer) for which the incriminated drugs have been prescribed | Case reported in VigiBase, APHP Entrepot de Données de Santé (EDS), Système National Des Données de Santé (SNDS) Databases and a retrospective international multicenter registry of ICI-associated myocarditis from inception to January 2025
Description of the population of patients having a cardio-vascular adverse event | Case reported in VigiBase, APHP Entrepot de Données de Santé (EDS), Système National Des Données de Santé (SNDS) Databases and a retrospective international multicenter registry of ICI-associated myocarditis from inception to January 2025
Cardio-vascular toxicity of ICIs. | Case reported in VigiBase, APHP Entrepot de Données de Santé (EDS), Système National Des Données de Santé (SNDS) Databases and a retrospective international multicenter registry of ICI-associated myocarditis from inception to January 2025
  Number of patients with cardiovascular adverse events with significant over-reporting ICIs
Description and added predictive value of electrocardiographic, echocardiographic, cardiac and muscle pathology, cardiac MRI and positron emission tomograph (PET) manifestations in patients with ICI associated myocarditis | Case reported in VigiBase, APHP Entrepot de Données de Santé (EDS), Système National Des Données de Santé (SNDS) Databases and a retrospective international multicenter registry of ICI-associated myocarditis from inception to January 2025
  Description and added predictive value of electrocardiographic, echocardiographic, cardiac and muscle pathology, cardiac MRI and positron emission tomograph (PET) manifestations in patients with ICI associated myocarditis

CONTACTS AND LOCATIONS:
Locations (1):
- AP-HP, Pitié-Salpêtrière Hospital, Department of Pharmacology, CIC-1421, Pharmacovigilance Unit, INSERM., Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moslehi JJ, Salem JE, Sosman JA, Lebrun-Vignes B, Johnson DB. Increased reporting of fatal immune checkpoint inhibitor-associated myocarditis. Lancet. 2018 Mar 10;391(10124):933. doi: 10.1016/S0140-6736(18)30533-6. No abstract available. PMID 29536852
- [Background] Salem JE, Manouchehri A, Moey M, Lebrun-Vignes B, Bastarache L, Pariente A, Gobert A, Spano JP, Balko JM, Bonaca MP, Roden DM, Johnson DB, Moslehi JJ. Cardiovascular toxicities associated with immune checkpoint inhibitors: an observational, retrospective, pharmacovigilance study. Lancet Oncol. 2018 Dec;19(12):1579-1589. doi: 10.1016/S1470-2045(18)30608-9. Epub 2018 Nov 12. PMID 30442497
- [Background] Salem JE, Allenbach Y, Vozy A, Brechot N, Johnson DB, Moslehi JJ, Kerneis M. Abatacept for Severe Immune Checkpoint Inhibitor-Associated Myocarditis. N Engl J Med. 2019 Jun 13;380(24):2377-2379. doi: 10.1056/NEJMc1901677. No abstract available. PMID 31189043
- [Background] Bonaca MP, Olenchock BA, Salem JE, Wiviott SD, Ederhy S, Cohen A, Stewart GC, Choueiri TK, Di Carli M, Allenbach Y, Kumbhani DJ, Heinzerling L, Amiri-Kordestani L, Lyon AR, Thavendiranathan P, Padera R, Lichtman A, Liu PP, Johnson DB, Moslehi J. Myocarditis in the Setting of Cancer Therapeutics: Proposed Case Definitions for Emerging Clinical Syndromes in Cardio-Oncology. Circulation. 2019 Jul 2;140(2):80-91. doi: 10.1161/CIRCULATIONAHA.118.034497. PMID 31390169
- [Derived] Power JR, Dolladille C, Ozbay B, Procureur A, Ederhy S, Palaskas NL, Lehmann LH, Cautela J, Courand PY, Hayek SS, Zhu H, Zaha VG, Cheng RK, Alexandre J, Roubille F, Baldassarre LA, Chen YC, Baik AH, Laufer-Perl M, Tamura Y, Asnani A, Francis S, Gaughan EM, Rainer PP, Bailly G, Flint D, Arangalage D, Cariou E, Florido R, Narezkina A, Liu Y, Sandhu S, Leong D, Issa N, Piriou N, Heinzerling L, Peretto G, Crusz SM, Akhter N, Levenson JE, Turker I, Eslami A, Fenioux C, Moliner P, Obeid M, Chan WT, Ewer SM, Kassaian SE, Johnson DB, Nohria A, Ben Zadok OI, Moslehi JJ, Salem JE; International ICI-Myocarditis Registry. Immune checkpoint inhibitor-associated myocarditis: a novel risk score. Eur Heart J. 2025 Jun 18:ehaf315. doi: 10.1093/eurheartj/ehaf315. Online ahead of print. PMID 40569849
- [Derived] Power JR, Dolladille C, Ozbay B, Procureur AM, Ederhy S, Palaskas NL, Lehmann LH, Cautela J, Courand PY, Hayek SS, Zhu H, Zaha VG, Cheng RK, Alexandre J, Roubille F, Baldassarre LA, Chen YC, Baik AH, Laufer-Perl M, Tamura Y, Asnani A, Francis S, Gaughan EM, Rainer PP, Bailly G, Flint D, Arangalage D, Cariou E, Florido R, Narezkina A, Liu Y, Sandhu S, Leong D, Issa N, Piriou N, Heinzerling L, Peretto G, Crusz SM, Akhter N, Levenson JE, Turker I, Eslami A, Fenioux C, Moliner P, Obeid M, Chan WT, Ewer SM, Kassaian SE; International ICI-Myocarditis Registry; Johnson DB, Nohria A, Zadok OIB, Moslehi JJ, Salem JE. Predictors and Risk Score for Immune Checkpoint-Inhibitor-Associated Myocarditis Severity. medRxiv [Preprint]. 2024 Jun 3:2024.06.02.24308336. doi: 10.1101/2024.06.02.24308336. PMID 38883792
- [Derived] Nguyen LS, Bretagne M, Arrondeau J, Zahr N, Ederhy S, Abbar B, Pinna B, Allenbach Y, Mira JP, Moslehi J, Rosenzwajg M, Salem JE. Reversal of immune-checkpoint inhibitor fulminant myocarditis using personalized-dose-adjusted abatacept and ruxolitinib: proof of concept. J Immunother Cancer. 2022 Apr;10(4):e004699. doi: 10.1136/jitc-2022-004699. PMID 35383117